CLINICAL TRIAL: NCT02604537
Title: Betamethason Versus Ketorolac Injection for the Treatment of DeQuervains Tenosynovitis
Brief Title: Betamethasone Versus Ketorolac Injection for the Treatment of DeQuervains Tenosynovitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15060
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: DeQuervain Tendinopathy
MeSH Terms: interventions — Betamethasone; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betamethasone (Active Comparator): 1 cc of 1% lidocaine (without epinephrine) plus 1 cc of 6 mg/ml betamethasone (Celestone)
  Interventions: Drug: betamethasone
- Ketorolac (Experimental): 1 cc of 1% lidocaine (without epinephrine) plus 1 cc of 30 mg/ml of ketorolac (Toradol)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: betamethasone — 1 cc of 1% lidocaine (without epinephrine) plus 1 cc of 6 mg/ml betamethasone
  Other Names: Celestone
  Arms: Betamethasone
Drug: Ketorolac — 1 cc of 1% lidocaine (without epinephrine) plus 1 cc of 30 mg/ml of ketorolac
  Other Names: Toradol
  Arms: Ketorolac

SUMMARY:
The purpose of this study is to determine if corticosteroid injection modifies the natural course of de Quervain tendinopathy compared to a toradol injection.

DETAILED DESCRIPTION:
If steroids are effective for Dequervain tenosynovitis because of their anti-inflammatory properties, then there is a reasonable and rational argument to be made for the local injection of NSAIDS (non-steroidal anti-inflammatory drugs) into the first dorsal extensor compartment. Ketorolac is an NSAID that has been proven efficacious in the treatment of another musculoskeletal condition. Moreover, compared to betamethasone (or other injectable corticosteroids), injection of ketorolac decreases the patient exposure to the potential side-effects of corticosteroids, especially that of elevation of blood sugar levels in diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DeQuervain tendinopathy
* Understands the local language and is willing and able to follow the requirements of the protocol
* Understands the informed consent and signs the institutional review board/independent ethics committee (IRB/IEC) approved informed consent form

Exclusion Criteria:

* Patients who have an allergy to lidocaine, celestone, or ketorolac, nonsteroidal anti-inflammatory drugs (NSAIDs), or acetylsalicylic acid (ASA)
* Patients who have an adverse reaction to lidocaine, celestone, or ketorolac (such as severe elevation of blood sugars in diabetics that caused medical complication)
* Patients who have received a prior steroid injection within the past three months
* Patients who have had a prior ipsilateral surgery for DeQuervain Tenosynovitis
* Patients that have a skin lesion at the location of injection (such as trauma, eczema, rash)
* Patients who have a current infection at the location of injection
* Patients who have had iontophoresis within three months
* Patients who are breast feeding, pregnant, or who plan to become pregnant in the next six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-10-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) of pain with finklestein test | 6 weeks post injection
  Visual Analog Scale (VAS) of pain measured on 0 (no pain) - 10 (worst possible pain)

SECONDARY OUTCOMES:
Visual analog scale (VAS) of pain with tenderness over tendon | pre injection, 2 weeks post injection, 6 weeks post injection
  Visual Analog Scale (VAS) of pain measured on 0 (no pain) - 10 (worst possible pain)
Visual analog scale (VAS) of pain on radial side of wrist | pre injection, 2 weeks post injection, 6 weeks post injection, 3 months post injection, 6 month post injection
  Visual Analog Scale (VAS) of pain measured on 0 (no pain) - 10 (worst possible pain)
The Disabilities of the Arm, Shoulder, and Hand Score (DASH) | pre injection, 2 weeks post injection, 6 weeks post injection, 3 months post injection, 6 months post injection
  Patient-reported evaluation of symptoms as well as ability to perform certain activities. Score is 0-100 (higher scores indicate greater disability). Must answer at least 27/30 questions. Score is 1 to 5 per question. Score is then summed and divided by the number of completed questions. subtract 1 from this number then multiply by 25.
Veterans-Rand 12 (VR-12) | pre injection, 2 weeks post injection, 6 weeks post injection, 3 months post injection, 6 months post injection
  Quality of life using VR-12 subscores. Physical Health (PCS) subscore and Mental Health (MCS) subscore, not summed. Range reported in weighted units. Both PCS/MCS are score 0-100 with 100 indicating the highest level of health.
Pinch Strength | pre-injection, 2 weeks post injection, 6 weeks post injection
Grip Strength | pre injection, 2 weeks post injection, 6 weeks post injection

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chadderdon, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States